CLINICAL TRIAL: NCT00027261
Title: A Phase I Trial to Evaluate the Safety, Tolerability and Immunogenicity of High-Dose Live Recombinant Canarypox ALVAC-HIV Vaccine (vCP1452) in Healthy, HIV-1 Uninfected Adult Participants
Brief Title: Safety and Immune Response Study of High-Dose Canarypox ALVAC-HIV Vaccine in Healthy, HIV Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 039; 10200 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2001-11-29; First posted 2001-11-30 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: Vaccines, Synthetic; HIV-1; AIDS Vaccines; CD8-Positive T-Lymphocytes; HIV Seronegativity; Avipoxvirus; Dose-Response Relationship, Immunologic; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: ALVAC(2)120(B,MN)GNP (vCP1452)

SUMMARY:
The purpose of this study is to see if the experimental vaccine, ALVAC-HIV (vCP1452) is safe and to study how the immune system responds to the vaccine. This trial is designed to determine whether a higher vaccine dose (6 times the usual dose) will elicit a higher immune response.

As of May 2001, over 200 people received the ALVAC-HIV (vCP1452) vaccine at the lower dose. The higher dose of the vaccine to be used in this study has not been given to humans previously. High doses of a similar vaccine have been given to a few people without serious side effects. In a recent study done in mice, higher doses of ALVAC-HIV produced stronger immune responses. It is possible that the doses of ALVAC-HIV given to humans are below the amount needed for the maximum immune response. Because the exact relationship between an increased immune response and its effectiveness in preventing HIV infection is uncertain, the HVTN will use the highest dose that can be manufactured.

DETAILED DESCRIPTION:
To date, adverse reactions to immunization with the various ALVAC-HIV candidate vaccines, including ALVAC-HIV (vCP1452), have been similar to those observed in healthy adults who have received other licensed vaccines of similar types. In a previous trial, even high doses of recombinant ALVAC vaccine were well tolerated in a group of participants that were significantly immunocompromised. In a recent study done in mice concerning dose escalation using the ALVAC-HIV vectors, the data demonstrated more robust immune responses with higher doses of ALVAC-HIV (vCP1452) in mice. It is certainly possible that the doses of ALVAC-HIV given to humans are well below the amount needed for a maximal cytotoxic T lymphocyte (CTL) response. As the predictive value of a CTL response is at present unknown with respect to its efficacy in preventing or ameliorating HIV acquisition or infection, the HVTN will utilize the highest dose that can be currently manufactured.

All study products are to be administered intramuscularly. Participants will receive 1 of 3 injections. Group A will receive a high dose of vaccine, group B will receive a low dose of vaccine, and group C will receive a placebo. Participants are inoculated at 4 time points. Assessment of product safety includes clinical observation, monitoring of hematological, chemical, and immunologic parameters, and a social harms questionnaire. Safety will be evaluated by monitoring of participants for local and systemic adverse reactions during the course of the trial. Participants will be monitored longitudinally for HIV-specific serologic and cellular immune responses.

ELIGIBILITY:
Inclusion Criteria

Participants may be eligible for this study if they:

* Are between the ages of 18 and 60.
* Are in good general health.
* Have a CD4 count of 400 or more cells/mm3.
* Do not have hepatitis C or active hepatitis B.
* Have had a negative HIV blood test within 8 weeks prior to enrollment.
* Use approved methods of contraception.
* Have access to a participating site and are available for follow-up for 18 months.
* Complete a questionnaire evaluating the participant's understanding of the study prior to enrollment.
* Give written informed consent.

Exclusion Criteria

Participants may not be eligible for this study if they:

* Are pregnant or breast-feeding.
* Have received a live vaccine within 30 days prior to enrollment.
* Have received a killed vaccine or allergy treatment with injections within 14 days prior to study vaccine.
* Have used experimental research agents within 30 days prior to enrollment.
* Have received HIV-1 vaccines or placebo in a previous HIV vaccine trial.
* Have received blood products 120 days before HIV screening.
* Have received immunoglobulin 60 days before HIV screening.
* Have a history of serious harmful reactions to vaccines.
* Have a history of disease of the immune system.
* Have a history of cancer, unless it has been surgically removed and in the estimate of the investigator is not likely to happen again during the study period.
* Are using or have used (within past 6 months) drugs that interfere with the immune system.
* Have a history of type I or type II diabetes.
* Have thyroid disease.
* Have unstable asthma.
* Are currently taking preventive anti-TB therapy.
* Have a seizure disorder.
* Have a bleeding disorder that was diagnosed by a physician.
* Have had their spleen removed.
* Have angioedema with serious episodes.
* Have active syphilis.
* Have hypertension.
* Have mental problems that would interfere with the protocol.
* Have any other problems that, in the judgment of the investigator, would interfere with the study.
* Have a body mass index less than 20.
* Are allergic or sensitive to egg products.
* Have active tuberculosis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Goepfert, Study Chair
Locations (13):
- United States (13):
  - Alabama Vaccine CRS, Birmingham, Alabama
  - San Francisco Vaccine and Prevention CRS, San Francisco, California
  - UCSF, Gen. Clinical Research Ctr., Mt. Zion Hosp., San Francisco, California
  - Project Brave HIV Vaccine CRS, Baltimore, Maryland
  - Brigham and Women's Hosp. CRS, Boston, Massachusetts
  - Fenway Community Health Clinical Research Site (FCHCRS), Boston, Massachusetts
  - Saint Louis Univ Health Sciences Ctr, St Louis, Missouri
  - NY Blood Ctr./Union Square CRS, New York, New York
  - Univ. of Rochester HVTN CRS, Rochester, New York
  - Miriam Hospital's HVTU, Providence, Rhode Island
  - Vanderbilt Vaccine CRS, Nashville, Tennessee
  - Infectious Diseases Physicians, Inc., Annandale, Virginia
  - FHCRC/UW Vaccine CRS, Seattle, Washington

REFERENCES:
- [Result] Goepfert PA, Horton H, McElrath MJ, Gurunathan S, Ferrari G, Tomaras GD, Montefiori DC, Allen M, Chiu YL, Spearman P, Fuchs JD, Koblin BA, Blattner WA, Frey S, Keefer MC, Baden LR, Corey L; NIAID HIV Vaccine Trials Network. High-dose recombinant Canarypox vaccine expressing HIV-1 protein, in seronegative human subjects. J Infect Dis. 2005 Oct 1;192(7):1249-59. doi: 10.1086/432915. Epub 2005 Aug 31. PMID 16136469